CLINICAL TRIAL: NCT05640141
Title: Pre-demential Motoric Cognitive Risk Syndrome in Ageing Subjects - Prediction of Cognitive Decline and Identification of Underlying Mechanisms
Brief Title: Pre-demential Motoric Cognitive Risk Syndrome in Ageing Subjects
Acronym: PRESAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: PRESAGE
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2021-12

CONDITIONS: Motoric Cognitive Risk Syndrome; Mild Cognitive Impairment; Alzheimer Disease; Dementia
Keywords: MRI; Cognition; Gait; Executive functions; Virtual reality; Motion capture
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — 24,25-oxidolanosterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Control group composed of 80 healthy aged volunteers.
  Interventions: Procedure: MRI evaluation; Behavioral: Actimetry & IMU; Behavioral: Gait evaluation; Behavioral: Neuropsychological evaluation
- Motoric Cognitive Syndrom: MCR group composed of 80 MCR participants.
  Interventions: Procedure: MRI evaluation; Behavioral: Actimetry & IMU; Behavioral: Gait evaluation; Behavioral: Neuropsychological evaluation

INTERVENTIONS:
Procedure: MRI evaluation — Multimodal MRI evaluation :
  * T1 structural,
  * Resting echo planar imaging
  * Diffusion-weighted imaging
  * Arterial sping labeling
  * Fluid-attenuated inversion recovery
Behavioral: Actimetry & IMU — Evaluation of daily activities and life rythms (physical activity, inactivity, sleep) using actimeters (Motion 8), inertial sensors (GaitUP) and questionaires during 14 days :
  * Actimetry : evaluation of daily activity and inactivity, sleep rythms
  * Inertial sensors : gait evaluation during daily activities
  * Questionaires : sleep (Spiegel & St Mary's Hospitral) and fatigue (MFI-20)
Behavioral: Gait evaluation — Evaluation of gait characteristics (spatio-temporal parameters & non-linear characteristics) in virtual environment :
  * Locomotor simple task : gait only in congruent environment
  * Locomotor dual task : gait in similar environment combined with a visually displayed Stroop task
  * Sensorimotor gait adaptaition : evaluation of the adaptation capability throughout a split-belt treadmill sequence (realized in simple or dual -combined with the visual Stroop task-)
Behavioral: Neuropsychological evaluation — Complete neuropsychological examination including attentional and executive functions, learning and retrieval abilities in episodic memory and general cognitive skills :
  * Divided attention (TAP; test of attentional performance)
  * California Verbal Learning Test
  * The Rey-Osterrieth Complex Figure
  * Symbol search and coding (WAIS-IV)
  * Go/No-go (TAP)
  * Flexibility (TAP)
  * Original task of multimodal integration
  * Verbal fluencies (GREFEX)

SUMMARY:
The main aim of the study is to characterize and understand the pathological mechanisms underlying the motoric cognitive risk syndrome, which is a predictor of Alzheimer disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is affecting more than 46.8 million people worldwide, making dementia one of the greatest public health challenges of the 21st century. The progression of AD is slow with a presymptomatic course over several years to decades, during which pathophysiological changes are underway, but the disease has not yet caused any noticeable symptoms to warrant a clinical diagnosis. A strong effort is ongoing to identify biomarkers preceding cognitive decline that can aid diagnosis and early intervention. Criteria for the motoric cognitive risk syndrome (MCR), including subjective cognitive decline (SCD) and slower preferred walking speed, but otherwise normal functioning, are powerful risk indicators of developing cognitive impairment and dementia. The presence of MCR is associated with a more than three-fold risk of developing dementia while the risk is only two-fold for SCD or slow gait alone. However, the pathophysiology of MCR is unknown and getting into the processes that cause such condition is needed to complement the MCR-based criteria and increase their predictive validity of cognitive decline and dementia. Impaired attentional control related to white matter alterations of presumed vascular origin may be responsible for the MCR phenotype. Individuals with SCD exhibit loss of white matter integrity in brain regions typically involved in attentional control, and abnormally slow gait has been linked to the disruption of white matter tracts associated with executive attention. Furthermore, a deeper understanding of MCR requires considering not only regional white matter changes but also the individuals' cognitive capacity to cope with brain damages, namely the cognitive reserve. Hence, the PRESAGE project intends to evaluate the interplay of white matter integrity and cognitive reserve on attentional control in MCR and non-MCR individuals aged 60 or older. Attentional control will be explored at both the behavioral and brain levels using dual-task challenges where individuals will have to divide attention between a cognitive (stroop) task and a motor task (walking). The working hypothesis is that the dual-task cost - a proxy of attentional control - is predictive of white matter abnormalities which, when adjusted for cognitive reserve, age and sex, should discriminate between MCR and non-MCR individuals. The project also includes a prospective, longitudinal study (two-year follow-up) whose purpose is to determine whether this marker, alone or in combination with other potentially relevant markers (i.e., neuropsychological, functional and chronobiological), have predictive value for conversion from MCR to mild cognitive impairment and dementia. Findings will increase knowledge about the pathophysiology of MCR and will contribute to improve MCR criteria and early identification of at-risk individuals.

ELIGIBILITY:
Inclusion criteria:

* Aged 55-75 years
* Right-handed as assessed by the Edinburgh Inventory
* Health Insurance
* Able to follow experimental instructions
* Consent
* Independent in daily life activities as assessed by Katz autonomy score, ADL and IADL

Inclusion criteria (MCR group specific)

* Reduced gait speed as assessed by the 4m or 10m walk test value compared to normative values (Bohannon & Williams Andrews, 2011)
* Subjective cognitive complaint as assessed by dedicated questionnaire
* Subnormal cognitive function as assessed by the Montreal Cognitive Assessment (MoCA) test with score > 23

Inclusion criteria (Controls group specific)

- Subnormal cognitive function as assessed by the Montreal Cognitive Assessment (MoCA) test with score > 23

Exclusion criteria:

* Uncorrected visual or auditive deficits not allowing the realization of the experiment
* Evolutive disease (such as cancer)
* Active depression
* Neurological or psychiatric antecedent
* Neuromuscular impairment
* BMI < 35
* Counter-indication to MRI

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Controls : health volunteers without any reduced gait speed or cognitive complaint MCR : reduced gait speed, cognitive complaint Both : normal cognitive function
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Prediction accuracy to detect MCR participants will be computed using Machine learning | Baseline
  Several machine learning algorithms will be used to tell apart healthy from MCR participants. These classification procedures will bring several metrics including prediction accuracy, sensitivity and specificity scores.

SECONDARY OUTCOMES:
MRI - Brain volumes | Baseline
  Grey and white matter atrophy, grey matter structural covariation and white matter hyperintensity will be assessed.
MRI - Connectivity | Baseline
  Brain connectivity (covariation patterns) in each group will be computed.
Gait - Dual task cost | Baseline
  Difference in spatio-temporal and non-linear gait parameters bewteen simple and dual task / between groups
Gait - Sensorimotor adaptation and savings | Baseline
  Difference in terms of sensorimotor adaptation on split-belt treadmill bewteen groups

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Denise, MD, PhD, Principal Investigator — CHU de Caen Normandie
Locations (1):
- CHU de Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided